CLINICAL TRIAL: NCT05184439
Title: Clinical, Radiological and Isokinetic Evaluation of Adductor Magnus Tenodesis in Patients With Recurrent Patellar Dislocation.
Brief Title: Evaluation of Adductor Magnus Tenodesis in Patients With Recurrent Patellar Dislocation.
Status: Completed | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-BCO.67/2021-A
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Patellar Dislocation; Patellar Instability; Patellofemoral Osteoarthritis
Keywords: Recurrent Patellar Dislocation; Patellar instability; Isokinetics; Adolescents
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group after surgery: 33 children and adolescents (39 knees) with recurrent patellar dislocation were treated with MPFL reconstruction using the adductor magnus tendon between 2010 and 2012. The group is under clinical observation with evaluation being made.
  Interventions: Procedure: Adductor magnus tenodesis for recurrent patellar dislocation

INTERVENTIONS:
Procedure: Adductor magnus tenodesis for recurrent patellar dislocation — In all 33 patients (39 knees) adductor magnus tenodesis was performed to stabilise the patella. Adductor magnus tendon was harvested, cut proximally and fixed to the patella with proper tension.

SUMMARY:
Between 2010 and 2012, 33 children and adolescents (39 knees) with recurrent patellar dislocation were treated with MPFL reconstruction using the adductor magnus tendon.The aim of the study is to assess the effectiveness of this surgical procedure in long follow-up. The outcomes will be evaluated functionally (Lysholm knee scale, the Kujala Anterior Knee Pain Scale, and isokinetic examination) and radiographically (Caton-Deschamps index, sulcus angle, congruence angle, and patellofemoral angle). This is a continuation of the research published in 2015 with longer follow-up at least 10 years. All available patients will be evaluated with the same protocol, using the same methods and devices. Functional outcome is planned to be measured with scales as above. In radiological assessment Merchant and lateral knee weight bearing view and additionally MRI will be performed. Isokinetic test will be performed in two speeds of 60 and 180 deg/s. Most of important isokinetic parameters such as peak torque, torque in 30 deg, time to peak torque, peak torque to body weight both for quadriceps and hamstrings will be measured and compared to those from former research. Dedicated statistical test will be used for both: analysis of present status and differences from former results.

DETAILED DESCRIPTION:
Recurrent dislocation of the patella is a common orthopaedic problem which occurs in about 44% of cases after first-time dislocation. In most cases of first-time patellar dislocation, the medial patellofemoral ligament (MPFL) becomes damaged. Between 2010 and 2012, 33 children and adolescents (39 knees) with recurrent patellar dislocation were treated with MPFL reconstruction using the adductor magnus tendon. The aim of the study is to assess the effectiveness of this surgical procedure in long follow-up. The outcomes will be evaluated functionally (Lysholm knee scale, the Kujala Anterior Knee Pain Scale, and isokinetic examination) and radiographically (Caton-Deschamps index, sulcus angle, congruence angle, and patellofemoral angle). This is a continuation of the research published in 2015 with longer follow-up at least 10 years. All available patients will be evaluated with the same protocol, using the same methods and devices. Functional outcome is planned to be measured with scales as above. In radiological assessment Merchant and lateral knee weight bearing view and additionally MRI will be performed. Isokinetic test will be performed in two speeds of 60 and 180 deg/s. Most of important isokinetic parameters such as peak torque, torque in 30 deg, time to peak torque, peak torque to body weight both for quadriceps and hamstrings will be measured and compared to those from former research. Dedicated statistical test will be used for both: analysis of present status and differences from former results.

ELIGIBILITY:
Inclusion Criteria:

* patellar dislocation that had occurred at least twice,
* positive apprehensive test,
* completed research protocol
* age under 18 years at the time of surgery (adductor magnus tenodesis according to Avikainen)

Exclusion Criteria:

* first-time patellar dislocation
* habitual patellar dislocation
* patients with osteochondral fracture

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population consists of 33 patients (39 knees operated) after abductor magnus tenodesis for recurrent patellar dislocation with age under 18 at the time of surgery. With follow-up at least 10 years, present age of the subjects between 15 and 27 years.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Apprehension test | up to six months
  Fear during patellar passive lateralisation
Lysholm Score | up to six months
  Subjective outcome evaluation scale
Kujala Score | up to six months
  Subjective outcome evaluation scale
Sulcus angle | up to six months
  Index describing trochlear shape
Congruence angle | up to six months
  Index describing patellar shift
Patellofemoral angle | up to six months
  Index describing patellar tilt
Caton-Deschamps index | up to six months
  Index describing patellar height
Peak torque | up to six months
  Isokinetic evaluation in speeds 60 and 180 degree per second, both for quadriceps and hamstrings, Units of Measure - Newton-Metre (Nm)
Torque in 30 deg | up to six months
  Isokinetic evaluation in speeds 60 and 180 degree per second, both for quadriceps and hamstrings, Units of Measure - Newton-Metre (Nm)
Time to peak torque | up to six months
  Isokinetic evaluation in speeds 60 and 180 degree per second, both for quadriceps and hamstrings, Units of Measure - seconds (s)
Peak torque to body weight | up to six months
  Isokinetic evaluation in speeds 60 and 180 degree per second, both for quadriceps and hamstrings, Units of Measure - Nm/kg

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Małecki, Ph.D., Study Director — Polish Mother Memorial Hospital Research Institute
Locations (1):
- Polish Mother Memorial Hospital Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
We will be ready to share our data upon reasonable request of other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2022-2030
Access Criteria: Upon reasonable request krzynormal@wp.pl